CLINICAL TRIAL: NCT03272087
Title: Rational Approach to Unilateral Pleural Effusion in Patients Suspected of Malignancy. Efficacy, Pain, Quality of Life, and Economy
Brief Title: Rational Approach to a Unilateral Pleural Effusion
Acronym: REPEAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patient inclusion cannot be completed within time limits
Sponsor: Naestved Hospital (Other)
Collaborators: University of Southern Denmark (Other); Odense University Hospital (Other); Zealand University Hospital (Other); University Hospital, Gentofte, Copenhagen (Other); Bispebjerg Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Simon Reuter, Ph.d.-Student, Naestved Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Resp-REPEAT-SIRE-2
Record Dates: First submitted 2015-11-05; First posted 2017-09-05 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Lung Neoplasms
Keywords: Thoracoscopy
MeSH Terms: conditions — Lung Neoplasms | interventions — Thoracoscopy; Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pleuroscopy (Active Comparator): According to BTS guideline thoracoscopy is the next procedure for patients who remain undiagnosed despite PET-CT and attempts to obtain biopsies. Eligible patients will be randomised to pleuroscopy or VATS. Patients with inconclusive pleuroscopy will proceed to VATS.
  Interventions: Device: Thoracoscopy
- VATS (thoracoscopy) (Active Comparator): According to BTS guideline thoracoscopy is the next procedure for patients who remain undiagnosed despite PET-CT and attempts to obtain biopsies. Eligible patients will be randomised to pleuroscopy or VATS. Patients with inconclusive pleuroscopy will proceed to VATS.
  Interventions: Device: VATS (thoracoscopy)

INTERVENTIONS:
Device: Thoracoscopy — 50 % of patients will have performed af medical thoracoscopy (pleuroscopy)
  Arms: Pleuroscopy
Device: VATS (thoracoscopy) — 50 % of patients will have performed a VATS (video-assisted thoracic surgery) thoracoscopy
  Arms: VATS (thoracoscopy)

SUMMARY:
Recurrent unilateral, non-infectious pleural exudate is suspicious for primary or secondary pleural malignancy. Both conditions are associated with 5-year survival of 10%. Work-up is difficult, as the pleural surface is large and <33% of pleural malignancies shed malignant cells to the pleural fluid. Even so, additional tissue biopsies are needed for establishing mutation status for targeted therapies.

Optimal imaging to guide tissue sampling is pivotal. PET-CT has higher sensitivity than conventional CT for detecting malignant lesions >10mm. However, no randomised trial has investigated differences in diagnostic accuracy, time-to-diagnosis, or economics. Falsely PET-positive lesions in e.g. colon, however, lead to more derived tests than do CT alone.

Gold standard for pleural tissue sampling is the surgical (VATS) thoracoscopy, allowing direct visual guiding of tissue sampling from all pleural surfaces. Yet, globally the medical (pleuroscopy) thoracoscopy is more widely used: cheaper, outpatient procedure, but allows only sampling from the parietal pleura. To date, no randomised studies have compared medical and surgical thoracoscopy concerning diagnostic hit rates, adverse events, or economics.

Investigators will perform two randomized studies to investigate whether

1. PET/CT is comparable to CT alone
2. VATS is comparable to pleuroscopy concerning hit rate, total investigations performed, time-to-diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with recurrent pleural effusion of unknown origin after a first pleural tap according to BTS guidelines.
2. Indication for thoracoscopy according to BTS guidelines.
3. Patients accept further investigation according to Danish and BTS guidelines.
4. Have received oral and written consent and agreed.
5. At the time of inclusion, above 18 years of age.

Exclusion Criteria:

1. Female patients: pregnancy or breastfeeding.
2. Lack of language comprehension.
3. Legally incompetent patients.
4. Life expectancy less than 3 month.
5. Contraindications to pleural tissue sampling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Number of patients diagnosed with cancer | 2 years
  (cancer = an unequivocal diagnosis of neoplastic disease; no cancer = clinically benign cause, and improved imaging at 6 month control).

SECONDARY OUTCOMES:
Quality of life | 1 month
  Questionnaire developed to assess the quality of life of cancer patients, QLQC 30
Total costs | 2 years
  calculated as costs patient-related, procedure-related, and overall
Pain | 2 years
  VAS scale
Quality of life | 1 month
  A standardised instrument for use as a measure of health outcome, EuroQol EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: Uffe Boedtger, MD, PhD, Study Director — Syddansk Universitet
Locations (1):
- Naestved Hospital, Næstved, Denmark